CLINICAL TRIAL: NCT00372840
Title: Efficacy and Feasibility of a Psychosocial Intervention Within the CCOP Context: Evaluation of the Facing Forward Guide to Facilitate Life After Active Cancer Treatment
Brief Title: Printed Education Materials in Patients Who Are Finishing Treatment for Stage I, Stage II, or Stage IIIA Breast Cancer, Colorectal Cancer, Prostate Cancer, or Chest Cancer
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Fox Chase Cancer Center (Other)
Collaborators: National Cancer Institute (NCI) (NIH)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Other
Other Study IDs: FCCC-FCRB-04-002-P; CDR0000464245 (Registry Identifier: PDQ (Physician Data Query)); NCI-2009-00569 (Registry Identifier: CTRP (Clinical Trials Reporting System)); 06-803 (Other: FCCC IRB)
Record Dates: First submitted 2006-09-06; First posted 2006-09-07 (Estimated); Last update posted 2020-03-02 (Actual); Status verified 2020-02

CONDITIONS: Breast Cancer; Colorectal Cancer; Lung Cancer; Malignant Mesothelioma; Prostate Cancer; Psychosocial Effects of Cancer and Its Treatment; Thymoma and Thymic Carcinoma
Keywords: psychosocial effects of cancer and its treatment; stage I breast cancer; stage II breast cancer; stage IIIA breast cancer; stage IIIA colon cancer; stage I prostate cancer; stage IIB prostate cancer; stage IIA prostate cancer; stage III prostate cancer; stage I non-small cell lung cancer; stage II non-small cell lung cancer; stage IIIA non-small cell lung cancer; limited stage small cell lung cancer; stage I rectal cancer; stage IIA rectal cancer; stage IIB rectal cancer; stage IIC rectal cancer; stage IIIA rectal cancer; pulmonary carcinoid tumor; stage I thymoma; stage II thymoma; stage III thymoma; stage I colon cancer; stage IIA colon cancer; stage IIB colon cancer; stage IIC colon cancer; stage IA malignant mesothelioma; stage IB malignant mesothelioma; stage II malignant mesothelioma; stage III malignant mesothelioma
MeSH Terms: conditions — Breast Neoplasms; Colorectal Neoplasms; Lung Neoplasms; Mesothelioma, Malignant; Prostatic Neoplasms; Thymoma; Colonic Neoplasms; Carcinoma, Non-Small-Cell Lung; Rectal Neoplasms | interventions — Early Intervention, Educational; Psychiatric Rehabilitation

ARMS (2):
- Arm I (Experimental): Patients receive a specific print intervention manual entitled Facing Forward Series: Life After Cancer Treatment and a general print intervention fact sheet entitled The Cancer Information Service, Questions and Answers.
  Interventions: Other: educational intervention
- Arm II (Active Comparator): Patients receive the general print intervention fact sheet entitled The Cancer Information Service, Questions and Answers.
  Interventions: Procedure: psychosocial assessment and care; Procedure: quality-of-life assessment

INTERVENTIONS:
Other: educational intervention
  Arms: Arm I
Procedure: psychosocial assessment and care
  Arms: Arm II
Procedure: quality-of-life assessment
  Arms: Arm II

SUMMARY:
RATIONALE: Printed educational materials, such as the Facing Forward Series: Life After Cancer Treatment manual, may help make the transition from cancer patient to cancer survivor easier in patients who are finishing treatment for cancer. It is not yet known if the Facing Forward Series: Life After Cancer Treatment manual and The Cancer Information Service, Questions and Answers fact sheet is more effective than the The Cancer Information Service, Questions and Answers fact sheet alone in helping to make life after cancer treatment easier and to improve quality of life in patients with breast cancer, colorectal cancer, prostate cancer, or chest cancer.

PURPOSE: This randomized clinical trial is studying how well printed education materials work in assisting patients who are finishing treatment for stage I, stage II, or stage IIIA breast cancer, colorectal cancer, prostate cancer, or chest cancer to make the transition from cancer patient to cancer survivor easier.

DETAILED DESCRIPTION:
OBJECTIVES:

Primary

* Determine the efficacy of a psychoeducational intervention comprising a specific print intervention manual (Facing Forward Series: Life After Cancer Treatment [Facing Forward manual]) and a general print intervention fact sheet (The Cancer Information Service, Questions and Answers) vs the general print intervention fact sheet only on the uptake of recommended actions (e.g., developing a wellness plan after treatment, dealing with pain and fatigue, finding support groups to deal with feelings after treatment, and dealing with family issues after treatment) in patients completing active treatment for stage I-IIIA breast, prostate, colorectal, or thoracic cancer.
* Explore patient process evaluations of the Facing Forward manual in terms of its usability, comprehension, and satisfaction.

Secondary

* Examine psychological outcomes (i.e., depressive symptoms, fear of recurrence, health-related quality of life, and self-efficacy) as a function of exposure to the Facing Forward manual.

OUTLINE: This is a multicenter, randomized, controlled, open-label, cohort study. Patients are stratified according to participating center, prior chemotherapy (yes vs no), and type of cancer (breast vs colorectal vs prostate vs thoracic). Patients are randomized to 1 of 2 arms.

* Arm I (intervention): Patients receive a specific print intervention manual entitled Facing Forward Series: Life After Cancer Treatment and a general print intervention fact sheet entitled The Cancer Information Service, Questions and Answers.
* Arm II (control): Patients receive the general print intervention fact sheet entitled The Cancer Information Service, Questions and Answers.

In both arms, patients are evaluated at baseline (within 18 days of the patient's final cancer treatment visit), 8 weeks (via mailed home materials), and then at 6 months (via mailed home materials). Baseline evaluations include background information (i.e., demographics and medical status), baseline use of educational materials, survivorship activities, and psychological factors (i.e., depressive symptoms, quality of life, fear of recurrence, and self-efficacy). Psychological factors are also reassessed at 8 weeks and 6 months, as well as use of educational materials and survivorship activities.

For patients in both arms, uptake of recommended actions are reassessed. Patients in arm I complete ratings of the Facing Forward Series: Life After Cancer Treatment manual usability, comprehension, and satisfaction at 8 weeks and 6 months.

PROJECTED ACCRUAL: A total of 332 patients will be accrued for this study.

ELIGIBILITY:
DISEASE CHARACTERISTICS:

* Diagnosis of breast, colorectal, prostate, or thoracic cancer*

  * Stage I-III disease
  * Approaching, attending, or already attended with the past 28 days, the last treatment appointment of chemotherapy and/or radiotherapy NOTE: *Stage IIIA disease for thoracic cancer and excluded mesothelioma; if small cell lung cancer is present must be limited stage disease
* No more than 1 primary cancer
* No recurrent disease
* Hormone receptor status not specified

PATIENT CHARACTERISTICS:

* Male or female
* Menopausal status not specified
* Able to speak/read English at an 8th grade level

PRIOR CONCURRENT THERAPY:

* See Disease Characteristics
* No prior brachytherapy only
* No prior surgery only (i.e., must have received prior adjuvant therapy and surgery)

Ages: 18 Years to 120 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 340 (Actual)
Dates: Start 2006-05; Primary Completion 2010-11 (Actual); Study Completion 2013-03 (Actual)

PRIMARY OUTCOMES:
Uptake of recommended actions | 18 days, 8 weeks, 6 months after completion of treatment
Number of sections of the Facing Forward manual read with satisfaction and comprehension | 18 days, 8 weeks, 6 months after completion of treatment

SECONDARY OUTCOMES:
Changes in psychological outcomes from baseline to 8-week follow-up | 8 weeks, 6 months after completion of treatment

CONTACTS AND LOCATIONS:
Overall Officials: Suzanne M. Miller, PhD, Principal Investigator — Fox Chase Cancer Center
Locations (1):
- Fox Chase Cancer Center - Philadelphia, Philadelphia, Pennsylvania, United States

REFERENCES:
- [Background] Green BL, Krupnick JL, Rowland JH, Epstein SA, Stockton P, Spertus I, Stern N. Trauma history as a predictor of psychologic symptoms in women with breast cancer. J Clin Oncol. 2000 Mar;18(5):1084-93. doi: 10.1200/JCO.2000.18.5.1084. PMID 10694561